CLINICAL TRIAL: NCT06256471
Title: The Impact of Parasitic Infection on the Course of Multiple Sclerosis and Nephrotic Syndrome
Brief Title: The Impact of Parasitic Infection on Multiple Sclerosis and Nephrotic Syndrome
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Monica Refaat Hakeem Saweries, Demonstrator, Assiut University
Other Study IDs: Parasitic infection
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Parasitic Disease
MeSH Terms: conditions — Parasitic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Follow up of multiple sclerotic and nephrotic syndrome patients after 3 months — Follow up of multiple sclerotic and nephrotic syndrome patients after 3 months for detection of impact of parasitic infection on these diseases courses

SUMMARY:
1. Detection of the prevalence of parasitic infections amoung patients with multiple sclerosis and nephrotic syndrome at Assiut University Hospitals.
2. Detection of the effect of parasitic infections on these diseases courses.
3. Inform authorities about the importance of management of parasitic infections in those patients.

DETAILED DESCRIPTION:
Parasitic protozoal infections have prominent immunomodulatory changes in different autoimmune diseases. Moreover, helminths and their derivatives were established to have a protective role. Clinical trials of autoimmune diseases have tested the obvious helminths' immunomodulatory effect in inflammatory bowel disease, multiple sclerosis and rheumatoid arthritis . Autoimmunity is the immune system's inability to differentiate between foreign and self-antigens, resulting in damage of the healthy tissues . Recently, strong epidemiological studies revealed a steady increase in autoimmune diseases incidence in the developed countries. Also, The prevalence of the autoimmune diseases varies between rural and urban areas within the same country . The high records of autoimmune diseases incidences in these countries is attributed to the decline in infectious diseases prevalence "hygiene hypothesis ".

Multiple sclerosis (MS) is an inflammatory demyelinating disease affecting the CNS. Although its etiology remains obscure, several lines of evidence show that autoimmunity has a major role in the disease pathogenesis . Recent researches explain that parasitic infections can alter the disease course . Which is in the form of decreased number of relapses, minimal change in disability scores and lower MRI activity .

Childhood nephrotic syndrome (NS) is a worldwide disease with incidence and prognosis vary greatly according to the geographic distribution, with a prevalence of 15 per 100 000 under 16 years of age and higher incidence in South Asian (Pakistani, Indian, and Bangladeshi) and Arab children . NS is considered as a disease with immune impairment, Also some infections are found to be related to nephrotic syndrome . Parasitic infections may possibly be nonspecific triggers of NS . For instance, parasitic infections have been known to be associated with immune complex- mediated glomerular lesions . Moreover, parasites can mediate Altered T-helper cell cytokine expression, binding of autoantibodies to glomerular autoantigens, and immune complex formation .

The present study clarifies two very interesting and yet unexplored potentials, Do parasitic infections aggravate or ameliorate the course of autoimmune diseases? Also, what is the prevalence of parasitic infections in MS and NS in our governorate?

ELIGIBILITY:
Inclusion Criteria:

- 1- clinically and laboratory-confirmed autoimmune diseases according to: multiple sclerosis attending Neurology Department at Assiut University Hospitals.

2- clinically and laboratory-confirmed autoimmune diseases according to: nephrotic syndrome attending Pediatric Department at Assiut University Hospitals.

Exclusion Criteria:

* Patients with other commodities especially which cause secondary immune deficiencies like diabetes mellitus, patients with chronic liver disease or kidney diseases other than NS, malignancies and pregnant females.

Max Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: clinically and laboratory-confirmed autoimmune diseases according to: multiple sclerosis attending Neurology Department at Assiut University Hospitals and clinically and laboratory-confirmed autoimmune diseases according to: nephrotic syndrome attending Pediatric Department at Assiut University Hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
The impact of parasitic infection on multiple sclerosis and nephrotic syndrome | Baseline
  Detection of prevalence of parasitic infection on multiple sclerosis and nephrotic syndrome and the effect of parasitic infection on these diseases courses

REFERENCES:
- [Background] Strachan DP. Hay fever, hygiene, and household size. BMJ. 1989 Nov 18;299(6710):1259-60. doi: 10.1136/bmj.299.6710.1259. No abstract available. PMID 2513902
- [Background] Correale J, Farez M. Association between parasite infection and immune responses in multiple sclerosis. Ann Neurol. 2007 Feb;61(2):97-108. doi: 10.1002/ana.21067. PMID 17230481